CLINICAL TRIAL: NCT07246499
Title: Characteristics of Transmucosal Abutments for Dental Implants.
Brief Title: Multicentre Study on the Impact of Transmucosal Abutment Surface Characteristics on Peri-implant Tissues.
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Collaborators: University of Santiago de Compostela (Other)
Responsible Party: Principal Investigator, Juan Carlos Bernabeu Mira, Professor, PhD., University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1. UV-INV_ETICA-3792382
Record Dates: First submitted 2025-11-17; First posted 2025-11-24 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-10

CONDITIONS: Peri-implant Tissue Healing Assessed by Proteomic Analysis
Keywords: peri-implant healing; proteomics; tissue regeneration; Evaluation of proteomic outcomes in peri-implant tissue healing.; Pink anodized implant abutment; Grey machined implant abutment

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pink anodized titanium implant abutment. (Experimental): Participants will receive a pink anodized implant abutment, and peri-implant tissue healing will be assessed through proteomic analysis.
  Interventions: Device: Pink anodized implant abutment.
- Grey machined titanium implant abutment. (Active Comparator): Participants will receive a grey machined implant abutment, and peri-implant tissue healing will be assessed through proteomic analysis.
  Interventions: Device: Grey machined implant abutment.

INTERVENTIONS:
Device: Pink anodized implant abutment. — Participants will receive a pink anodized titanium implant abutment placed during the surgical and osseointegrated phase of treatment. Peri-implant tissue healing will be assessed over a three-month follow-up period through clinical examination and proteomic analysis.
  Other Names: Pink anodized dental abutment; Anodized titanium abutment
  Arms: Pink anodized titanium implant abutment.
Device: Grey machined implant abutment. — Participants will receive a grey machined titanium implant abutment placed during the surgical and osseointegrated phase of treatment. Peri-implant tissue healing will be assessed over a three-month follow-up period through clinical examination and proteomic analysis.
  Other Names: Grey machined dental abutment; Machined titanium abutment
  Arms: Grey machined titanium implant abutment.

SUMMARY:
The main objective of the study is to perform proteomic adsorption analysis on machined (grey) and anodised (pink) surfaces and compared them. The aim is to evaluate the regenerative potential involving improvement in the healing of peri-implant soft tissues in patients with dental implants. This surgery is indicated in healthy patients when they lost their teeth.

The main question it seeks to answer is:

- In dental abutments, is anodised surface more effective than machined surface in terms of the degree of healing?

The study will include patients who need this type of surgery and meet specific clinical criteria. Each patient will have one of the two dental abutments applied as part of the standard surgical procedure. Subsequently, participants will undergo clinical and proteomic follow-up assessments to evaluate the progress and extent of peri-implant tissue healing over a three-months period.

ELIGIBILITY:
Inclusion Criteria:

* Number of missing teeth and, therefore, number of implants required.
* A minimum of 4 implants, either single or bridges, must always be used in order to place 2 machined abutments and 2 anodised abutments.
* Sufficient bone dimensions for a minimum implant diameter of 3.5-4 mm and length of 6-8 mm, without prior bone regeneration.
* Patients who require indirect breast lift simultaneously with implant placement may be included in the study.
* Minimum keratinised mucosa dimension of 1.5-2.0 mm in all directions.
* Previous healthy bone condition for 3 months without infection.
* Periodontal health with no history of periodontitis (Silness and Löe plaque index, bleeding on probing (BOP) < 3 mm).

Exclusion Criteria:

* Patients unable to complete follow- up.
* Implant failures.
* Contamination of the sample during transfer from the abutment to the test tube.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Proteomic analysis of peri-implant tissue healing. | 7 days and 3 months after abutment placement.
  Proteomic profiling of peri-implant tissues will be performed to characterise protein expression patterns associated with tissue healing, enabling the identification of molecular markers of tissue regeneration.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The sharing of individual participant data is under consideration. Should data be shared in the future, all institutional regulations will be followed to protect participant confidentiality.